CLINICAL TRIAL: NCT03711292
Title: Using Behavioral Science to Reduce Inappropriate Antibiotic Use in Acute Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 31429-01; UL1TR001881 (NIH)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2018-10

CONDITIONS: Antimicrobial Stewardship; Acute Bronchitis; Upper Respiratory Infection
Keywords: Emergency Department; Urgent Care Center; Behavioral Sciences
MeSH Terms: conditions — Bronchitis; Respiratory Tract Infections; Emergencies | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped Wedge Cluster Randomized (Experimental): Antibiotic stewardship intervention
  Interventions: Behavioral: Antibiotic Stewardship

INTERVENTIONS:
Behavioral: Antibiotic Stewardship — For the 12-month intervention period, in a stepped-wedge fashion, sites will be exposed to a site-adapted multifaceted stewardship intervention consistent with CDC core elements for outpatient antimicrobial stewardship: commitment, action, monitoring, reporting and education, and also included a behavioral component that used individualized audit and feedback, peer comparison, and public commitment, in addition to standard patient and clinician education on antibiotic prescribing for antibiotic nonresponsive ARIs.

SUMMARY:
Stepped wedge behavioral intervention clinical trial looking at the impact of an antibiotic stewardship intervention on provider prescribing behavior for acute respiratory infections (ARIs), where the intervention is administered at the emergency department or urgent care center site level, using a cluster randomization process. Thus, every site and every provider are eligible to be exposed to the stewardship intervention, the cluster randomized stepped wedge process simply randomizes when they will be exposed. The overall study hypothesis is that providers will prescribe fewer unnecessary antibiotics to patients with ARIs after the intervention.

DETAILED DESCRIPTION:
Hypothesis: The primary hypothesis is that acute care ambulatory settings randomized to receive behavioral economic stewardship interventions will have decreased antibiotic prescribing rates for non-antibiotic appropriate ARIs, compared to contemporaneous antibiotic prescribing rates for non-antibiotic appropriate ARIs among control practices. This hypothesis will be evaluated in a linear mixed effects model will be used to estimate and test the group effect using group and time as fixed effects and practice site and provider as random effects. The interaction between time and group will be included to estimate and test the different group effect over time.

Design: The investigators will conduct a stepped wedge cluster randomized trial of acute care ambulatory visits to emergency departments and urgent care centers in a predominantly non-academic public hospital system. Clustering (by site) helps prevent treatment contamination between individual clinicians within the same site. The stepped wedge design will allow studying the effects of a complex intervention rolled out through a system over time, as often happens in the real-world, where State and Federal public health as well as site-based organization quality improvement interventions may be occurring at different times.

Treatment Assignment Procedures: For the 12-month intervention period, in a stepped-wedge fashion, sites will be exposed to a site-adapted multifaceted stewardship intervention consistent with Centers for Disease Control and Prevention (CDC) core elements for outpatient antimicrobial stewardship: commitment, action, monitoring, reporting and education, and also included a behavioral component that used individualized audit and feedback, peer comparison, and public commitment, in addition to standard patient and clinician education on antibiotic prescribing for antibiotic nonresponsive ARIs.

ELIGIBILITY:
The primary research subjects involved in this trial are prescribing providers who will be recruited from multiple clinical sites in Los Angeles County Department of Health Services.

Eligibility (provider)

Inclusion Criteria:

* Prescribing provider in an adult emergency department or urgent care center in the Los Angeles County Department of Health Services.

Exclusion Criteria:

* Provider has not treated a patient with an ARI

Eligibility (patient)

Inclusion Criteria:

* Treated at a Los Angeles County Department of Health Services facility with an ARI diagnosis
* Cared for by a provider and in practice site enrolled in the study
* Visit occurred during the 12-month intervention period, or the 12-month historical baseline period
* Did not have a visit with any ARI diagnosis in the prior 30 days

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing | 12 months
  The primary outcome measure is the rate of antibiotic prescribing for non-antibiotic-appropriate acute respiratory infections or in other words, acute respiratory infections that are presumed to be viral in nature. The International Classification of Diseases (ICD)-10 codes for primary outcomes are defined in detail in the clinical trials protocol document. These outcomes are computable clinical quality measures from the electronic health record. These are widely used in medicine to evaluate quality improvement and reliability and validity are generally supported.
  Visits are excluded from the primary analysis when: 1) patients have certain medical co-morbidities that make ARI guidelines less likely to apply, 2) patients had concomitant visit diagnoses indicating a non-ARI possible bacterial infection, or 3) patients had concomitant visit diagnoses indicating potentially antibiotic appropriate ARI diagnoses or other ARI diagnoses suggestive of a bacterial infection.

SECONDARY OUTCOMES:
Diagnostic drift | 12 months
  Throughout the course of the study, the investigators will also be monitoring "diagnostic drift" that may result in provider shifting diagnosis to avoid guideline conflicts that might trigger poor performance reports. An auditing program will measure diagnostic deviation from each clinician's historical rates of diagnosing acute respiratory infections.

CONTACTS AND LOCATIONS:
Overall Officials: Kabir Yadav, MDCM MS MSHS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Department of Health Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No